CLINICAL TRIAL: NCT05074914
Title: Mechanisms and Treatment of Unintentional Weight Loss After Oesophagectomy With Curative Intent
Brief Title: Unintentional Weight Loss After Oesophagectomy
Acronym: UWL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UWL-01
Record Dates: First submitted 2021-07-15; First posted 2021-10-12 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adenocarcinoma of the oesophagus (Experimental): curative oesophagectomy
  Interventions: Procedure: oesophagectomy
- Barrett's oesophagus (No Intervention): Weight stable patient under survelliance with Barrett's oespophagus

INTERVENTIONS:
Procedure: oesophagectomy — removal of oesophagus
  Arms: Adenocarcinoma of the oesophagus

SUMMARY:
The incidence of cancer of the oesophagus is increasing. While surgical removal of the tumour (oesophagectomy) may offer the best chance of cure, such major operations are associated with long-term complications such as poor appetite, unintentional weight loss and nutritional impairments. In the long-term, unintentional weight loss of 10-30% increases the risk of disease and death. However, a knowledge gap exists as there has been no comprehensive assessment of how this surgery changes the mechanisms of how the gut communicates with the brain (gut-brain pathways) and its relation to food intake and eating behaviour.

The aims of this study are to test the hypotheses that:

1. Oesophagectomy induces changes in the small intestine barrier (gut mucosa) and changes in hormonal signals after food consumption.
2. Oesophagectomy reduces appetite, eating behaviour, and food intake and shifts food selection from high-fat and high-glycaemic index items (quickly digested carbohydrates) to low-fat and low-glycaemic index items (slowly digested).

DETAILED DESCRIPTION:
Oesophageal cancer accounts for 27,700 deaths per year in the European Union (1). Oesophagectomy is a key component of state of the art multi-modal (preoperative chemo[radio] therapy) treatment for these patients (2).

Patients may require additional chemo(radio)therapy and/ or a feeding jejunostomy for the initial period after surgery. Half of the patients remain cancer free five years after oesophagectomy (3), however many of them have unintentional weight loss as the patients involuntarily reduce food intake (4).

Prior to curative surgery, unintentional weight loss is a common presenting feature among patients with oesophageal cancer. Initially after surgery, reduced food intake may be compounded by the impact of the operation on the patient. This can be due to inflammation of the gut mucosa during chemo(radio)therapy. However, in contrast to many other operations of similar complexity, when patients recover from the surgical insult and are cured of cancer, restoration of normal food intake does not typically occur (5).

Unintentional weight loss of 10-30% (from starting weight following surgery) increases long term morbidity and mortality even in those in remission of cancer. Effective nutritional support reduces early postoperative associated morbidity but does not modify long-term oncologic outcome even when surgical techniques, tumour size, and malignant potential are standardized. Empirical support that it is possible for patients to increase their food intake voluntarily after oesophagectomy remains equivocal. The investigators don't understand why these patients, who are tumour free, suffer unintentional weight loss (4).

The existing putative aetiological factors do not fully explain continued unintentional weight loss. Initially after surgery gastric emptying is delayed, but after 6 months gastric emptying is rapid. Pancreatic exocrine insufficiency and/or small intestinal bacterial overgrowth are present in 40% of patients after oespohagectomy. A subset of patients also experiences early postprandial intestinal discomfort (dumping syndrome) after consuming refined carbohydrates. However, the severity of bacterial overgrowth, pancreatic exocrine insufficiency, or dumping syndrome does not correlate with unintentional weight loss. Moreover, treatments of these do not consistently lead to weight regain. Another potential factor, the reduction of the "hunger hormone" ghrelin after oesophagectomy does not fully explain unintentional weight loss as ghrelin recovers to baseline levels after 12-24 month and therapy with ghrelin analogues has had limited success in terms of increasing long term food intake and bodyweight. Consequently, a knowledge gap exists as to which other factors involved in the gut-brain pathway are key to the profound degree of weight loss.

The investigators will conduct a series of experiments investigating the gut, eating behaviour, and food intake in 48 patients who will be recruited from the INCOGC. These patients are all eligible for treatment with curative intent involving removal of the food pipe tumor. As a comparator group, the investigators will also recruit 16 weight stable patients under surveillance for Barrett's oesophagus (a condition that can develop into cancer in a small number of people) in the Irish National Centre for Early Upper GI Neoplasia. The study visits will be time-matched and balanced for risk-factor profile, age and gender; the comparator group will confirm that, in the absence of surgery, all end-points are temporally stable. Each subject will be studied four times. Subjects will be excluded if cancer recurrence or ongoing therapy compromises the study protocol.

All patients before and after oesophagectomy have routine endoscopy (procedure to allow examination of the food pipe) as part of standard care which will allow us to easily conduct aim 1 as fresh tissue samples from the gut will be easily obtained during this routine investigation. The initial biopsy sample (pre-intervention) will be obtained during the surgical episode in theatre so that no additional endoscopies will be required. Aim 2 is conducted on a separate day as subjects will arrive in the Clinical Research Facility after an overnight fast (water allowed). Upon arrival on each test day, weight and height will be recorded and body composition will be assessed. Subjects will be given a standard 400 kcal meal and have serial blood tests 30 minutes apart. The progressive ratio task (a simple test in which an increasing number of computer mouse clicks is needed to earn a sweet) will be conducted followed by a buffet lunch and blood and stool test. In the early afternoon subjects are allowed to go home.

Biopsies, blood and stool samples will be collected. The investigators will correlate changes in gut cells, hormones and microorganisms with changes in food preferences and eating behaviour.

ELIGIBILITY:
Inclusion Criteria:

A. Oesophageal adenocarcinoma group:

* Planned for oesophagectomy with gastric conduit reconstruction
* Recurrence-free at least 12 months post-operatively
* Weight loss ≥10% from premorbid weight or require ongoing caloric supplementation

B. Barrett's oesophagus group:

-Barrett's oesophagus group who are under surveillance from INCEUGIN

Exclusion Criteria:

* Pregnant or breastfeeding, or planning to become pregnant
* Unable to swallow or need frequent dilatations ("stretches")
* Unable to eat semisolid food
* Allergies or dietary intolerance
* Diabetes mellitus type 1
* Reoccurrence of disease after surgery or are having another active form of cancer
* Taking medication which may impact gut hormone physiology
* Unstable cardiovascular disease
* A significant neurological condition
* A previous upper gastrointestinal resection
* A medical condition that would limit the ability to take part, that might impact certain test results or might make it unsafe for the patient to take these treatments.
* Difficulty reading, understanding or remembering the information we have given.
* Previous abdominal surgery.
* Treatment with GLP-1 receptor agonists or DPP-IV inhibitor or insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of the change in appetitive behaviour from baseline (before oesophagectomy) until 2 years following oesophagectomy using a progressive ratio task. | 0, 6, 12 and 24 months
  measured using Progressive ratio task
Direct measurement of changes in food intake from baseline (before oesophagectomy) until two years postoperatively using a standard buffet meal and weighing the specific foods before and after consumption. | 0, 6, 12 and 24 months
  weighted measurement of food consumed before and after eating
Direct measurement of changes in food selection from baseline (before oesophagectomy) until two years postoperatively using a standard buffet meal and observing the specific foods selection before and after consumption. | 0, 6, 12 and 24 months
  observed measurement of food selection before and after eating
Measurement of the change in postprandial gut hormone profiles from baseline (before oesophagectomy) until two years following oesophagectomy. | Every 30 minutes over a two hour period at 0, 6, 12 and 24 months
  Measured through plasma hormone levels taken before and after food consumption
Measurement of the change in plasma bile acid profiles from baseline (before oesophagectomy) until two years following oesophagectomy. | Every 30 minutes over a two hour period at 0, 6, 12 and 24 months
  Measured through plasma bile levels taken before and after food consumption
Measurement of the change in faecal gut microbiota from baseline (before oesophagectomy) until two years following oesophagectomy. | Every 30 minutes over a two hour period at 0, 6, 12 and 24 months
  Measured through stool samples and observation of changes to bacteria present
Quantification of changes in enteroendocrine cells in the mucosa of the proximal small bowel at baseline (before oesophagectomy) until 2 years postoperatively. | Baseline and up to 24 months postoperatively
  Measured through biopsy
Quantification of changes in gut microbiota in the mucosa of the proximal small bowel at baseline before oesophagectomy until 2 years postoperatively. | Baseline and up to 24 months postoperatively
  Measured through biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Carel Le Roux, Pr, MD, Study Chair — University College Dublin
Locations (1):
- St James University Hospital Clinical Research Centre, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stahl M, Mariette C, Haustermans K, Cervantes A, Arnold D; ESMO Guidelines Working Group. Oesophageal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi51-6. doi: 10.1093/annonc/mdt342. No abstract available. PMID 24078662
- [Background] Wilke TJ, Bhirud AR, Lin C. A review of the impact of preoperative chemoradiotherapy on outcome and postoperative complications in esophageal cancer patients. Am J Clin Oncol. 2015 Aug;38(4):415-21. doi: 10.1097/COC.0000000000000021. PMID 24351783
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] Baker M, Halliday V, Williams RN, Bowrey DJ. A systematic review of the nutritional consequences of esophagectomy. Clin Nutr. 2016 Oct;35(5):987-94. doi: 10.1016/j.clnu.2015.08.010. Epub 2015 Sep 12. PMID 26411750
- [Background] Martin L, Lagergren P. Long-term weight change after oesophageal cancer surgery. Br J Surg. 2009 Nov;96(11):1308-14. doi: 10.1002/bjs.6723. PMID 19847871